CLINICAL TRIAL: NCT05504083
Title: A Multicenter Randomized and Controlled Phase IIb Study to Evaluate the Efficacy and Safety of D-0120 Tablets in Patients with Primary Hyperuricemia
Brief Title: Evaluate the Efficacy and Safety of D-0120 in Primary Hyperuricemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0120-206
Record Dates: First submitted 2022-08-11; First posted 2022-08-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Benzbromarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- D-0120 group 1 (Experimental): take D-0120 dose 1 orally during the treatment period.
  Interventions: Drug: D-0120
- D-0120 group 2 (Experimental): take D-0120 dose 2 orally during the treatment period.
  Interventions: Drug: D-0120
- Benzbromarone (Active Comparator): take benzbromarone orally during the treatment period.
  Interventions: Drug: Benzbromarone
- D-0120 group 3 (Experimental): take D-0120 dose 3 orally during the treatment period.
  Interventions: Drug: D-0120

INTERVENTIONS:
Drug: D-0120 — Part A: Randomized in a 1:1:1 ratio through the randomization system, and assigned to D-0120 group 1, D-0120 group 2 or benzbromarone control group. Part B: Subjects will be assigned to D-0120 group 3.
  Arms: D-0120 group 1; D-0120 group 2; D-0120 group 3
Drug: Benzbromarone — Part A: Randomized in a 1:1:1 ratio through the randomization system, and assigned to D-0120 group 1, D-0120 group 2 or benzbromarone control group.
  Arms: Benzbromarone

SUMMARY:
This is a randomized, open-label, parallel-controlled, multicenter clinical trial in primary hyperuricemia patients with or without gout.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily takes part in the study after being fully informed,signs a written ICF, and agrees to follow procedures specified in the study protocol;
2. Subject who meets one of the following criteria:

   i. History of gout attack: Meeting 2015 ACR/EULAR Gout Classification Criteria and fasting serum uric acid ≥ 480 μmol/L at screening (local laboratory of study site) ii. For asymptomatic hyperuricemia, it is acceptable to meet either of the two criteria:
   1. Serum uric acid ≥ 420 μmol/L for at least 3 months (subject to hospital medical record or test report), diagnosis with hyperuricemia before screening, and fasting serum uric acid at screening ≥ 540 μmol/L (local laboratory of study site);
   2. Serum uric acid ≥ 420 μmol/L for at least 3 months (subject to hospital medical record or test report), diagnosis with hyperuricemia before screening, and fasting serum uric acid at screening ≥ 480 μmol/L (local laboratory of study site), with concomitant primary hypertension or primary hyperlipidemia or type 2 diabetes mellitus, which is treated with a stable dose of antihypertensive or lipid-lowering or hypoglycemic treatment for at least 3 months;
3. At screening, 18.0 kg/m2 ≤ body mass index (BMI) ≤ 32.0 kg/m2;
4. Hematology, Blood chemistry and Urinalysis examination were basically normal.

Exclusion Criteria:

1. Prior intolerance to benzbromarone or contraindication to medication;
2. Secondary hyperuricemia caused by tumor, chronic kidney disease, blood disease or drugs, etc.;
3. Arthropathy caused by arthritis rheumatoid, purulent arthritis, traumatic arthritis, psoriatic arthritis, pseudogout or systemic lupus erythematosus, etc.;
4. Arthropathy caused by chemotherapy, radiotherapy or chronic lead poisoning;
5. Urinary calculi confirmed by B-ultrasound during screening period;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with serum uric acid ≤ 360 μmol/L | Day 1 - Day 85
  Percentage of subjects with serum uric acid ≤ 360 μmol/L at week 12 of treatment - based on test results by the central lab.

SECONDARY OUTCOMES:
Percentage of subjects with serum uric acid≤ 360 μmol/L | Day 1 -Day 56
  Percentage of subjects with serum uric acid ≤ 360 μmol/L at weeks 4 and 8 of treatment - based on test results by the central lab;
Changes in serum uric acid | Day 1 - Day 85
  Changes in serum uric acid from baseline at weeks 4, 8 and 12 of treatment - based on test results by the central lab;
Change percentage in serum uric acid | Day 1 - Day 85
  Change percentage in serum uric acid from baseline at weeks 4, 8 and 12 of treatment - based on test results by the central lab.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (24):
- China (24):
  - Inner Mongolia Baogang Hospital, Baotou
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First People's Hospital of Changzhou, Changzhou
  - Foshan Nanhai People's Hospital, Foshan
  - Guangzhou First People's Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - The Second People's Hospital of Guangdong Province, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital Of University Of South China, Hengyang
  - Huzhou Third People's Hospital, Huzhou
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Gulou Hospital Affiliated to Nanjing University Gulou Hospital Affiliated to Nanjing University, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Ningbo
  - Changhai Hospital of Shanghai, Shanghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Qinghai Province People's Hospital, Xining
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zigong Fourth People's Hospital, Zigong